CLINICAL TRIAL: NCT01277484
Title: Single Arm, Open Label, Phase I Study for Dose and Schedule Finding of Decitabine in Patients With Higher-risk MDS and MDS/AML Receiving Allogeneic Stem Cell Transplantation
Brief Title: Dose Finding Study of Post-BMT Decitabine Maintenance Treatment in Higher-risk MDS and MDS/AML
Acronym: PODAC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Yoo-Jin Kim, Associate Professor, Seoul St. Mary's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEC-KOR-9007
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: decitabine; dose; schedule; safety; allogeneic stem cell transplantation
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decitabine, MDS treatment, IV injection (Experimental): For the patients who achieve remission after allogeneic BMT and meet the enrollment criteria, decitabine will be given at a dose of 5mg/kg/day ~ 15mg/kg/day iv over 1 hour for 5 consecutive days starting 42-90 days after transplantation. The drug will be repeated every 4 weeks for up to 12 cycles.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 1. Dose finding study (cycle 1-cycle4)
  * Indicated dose for 5 consecutive days every 28 days
  * Cohort 1: 5mg/m2 of decitabine
  * Cohort 2 and 3:Dose escalation up to 15mg/m2 using a mechanism-based pharmacokinetic / pharmacodynamic model
  Other Names: Dacogen

SUMMARY:
Brief Scientific Rationale:

Decitabine has been shown to be effective for treatment of MDS and associated with very limited extramedullary toxicity at the lower doses. Furthermore, the hypomethylating effects of decitabine require an extended period of therapy and are likely to be more beneficial in the setting of a minimal residual disease after transplantation. The drug might exert a cytoreductive effect on the MDS clone, but ex vivo expansion strategy using decitabine and HDAC inhibitor provides a potential to expand the number of hematopoietic stem cells. There are lots of evidence which showed the the drug have immunostimulatory effects and can be used to enhance graft-versus leukemia effects. And also, some investigator suggested that decitabine could induce FOXP3 expression, promoting the conversion of naïve T cells to Tregs which are known to suppress GVHD while maintaining GVL effect in allo-SCT setting. As such, decitabine is an ideal agent to be investigated in the post-transplant setting.

The investigators hypothesized that post-transplant maintenance therapy with decitabine may reduce relapse rate, which may maximize the beneficial effects from reduced TRM of ATG-containing FB4 or FB2 conditioning regimen in higher-risk MDS or AML evolving from MDS patients.

DETAILED DESCRIPTION:
1. Transplant course

   * BMT from an HLA-matched sibling or a suitably matched (up to 2-allele mismatched) family or unrelated donor will be performed according to the policies of the institute.
   * A preparative regimen will be started 6 days before the day of stem cell infusion

     1. Myeloablative-intensity conditioning regimen: FB4+ATG
     2. Reduced-intensity conditioning regimen; FB2+ATG
     3. Graft-versus-host disease prophylaxis
   * Sibling transplant: Cyclosporine and short-course Methotrexate
   * Unrelated transplant: Tacrolimus and short-course Methotrexate
   * The dose of calcineurin inhibitors (cyclosporine and tacrolimus) will be gradually tapered from day 60 (for all sibling transplants) or day 90 (for all unrelated transplants) and discontinued within 2 or 3 months after SCT in the absence of graft-versus-host disease.
2. Decitabine maintenance course

   * For the patients who finish the above transplant procedure and meet the enrollment criteria, decitabine will be given at a dose of 5mg/m2/day ~ 15mg/m2/day iv over 1 hour for 5 consecutive days. The drug will be repeated every 4 weeks for up to 12 cycles.
   * Dose escalation strategy between cohorts and between cycles in the same cohort patients will be based upon the quantitatively measured hematological toxicity (e.g., ANC or platelet count at nadir). In other words, a mechanism-based pharmacokinetic / pharmacodynamic model developed using sparsely sampled patients' PK data and toxicity response will be used to titrate next cycle doses for the patients and initial doses for new cohort patients. In other words, a mechanism-based pharmacokinetic / pharmacodynamic model developed using sparsely sampled patients' PK data and toxicity response will be used to titrate next cycle doses for the patients and initial doses for new cohort patients.

ELIGIBILITY:
Inclusion Criteria for allogeneic transplantation::

* Patients with a diagnosis of MDS (IPSS intermediate-2 or higher) before allogeneic transplantation
* HLA-compatible unrelated (HLA-A, -B, -C and -DRB1 matched or with 2 allele mismatch)
* Performance status < ECOG 2
* Acceptable organ function defined as:Serum creatinine < 1.5 times the institutional ULN,Serum bilirubin < 1.5 times the institutional ULN,AST, ALT and alkaline phosphatase < 3 times the institutional ULN.

Inclusion Criteria for decitabine maintenance therapy:

* 6 to 10 weeks after alloHSCT
* patients who are confirmed complete remission(CR) within 2 weeks for treatment start(CR:less than 5% blasts in an aspirate bone marrow sample or no leukemic blasts in the peripheral blood, no cytogenetic aberrations)
* Performance status < ECOG 2
* Acceptable organ function defined as:Serum creatinine < 1.5 times the institutional ULN,Serum bilirubin < 1.5 times the institutional ULN,AST, ALT and alkaline phosphatase < 3 times the institutional ULN.
* Platelet count ≥ 30,000/μL without platelet transfusion for 7 days and ANC ≥ 1,000/μL without colony stimulating factor support at the time of enrollment
* Written informed consent form

Exclusion Criteria:

* HIV positive
* Active uncontrolled infection
* Pregnancy or breastfeeding
* patients who have residual disease after allo SCT or primary graft failure
* Uncontrolled grade 3- 4 acute GVHD
* patients who are known or suspected hypersensitivity to decitabine
* patient who are not suitable for the trial in accordance with principal investigator's decision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2014-09 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Dose and schedule finding of post-BMT Decitabine Treatment | For up to 2 years after the start of Decitabine
  To find the safe dose and schedule of administration of the drug decitabine that can be given to patients with higher risk MDS or secondary AML evolving from MDS who received allogeneic stem cell transplantation

SECONDARY OUTCOMES:
Transplant outcomes of Decitabine maintenance treatment following transplantation | For up to 2 years after the start of Decitabine
  To evaluate the benefit of maintenance therapy with decitabine in prolonging the duration of survival and relapse-free survival after allo-SCT.
  To evaluate the effect of maintenance therapy with decitabine on donor chimerism,GVHD, and other transplant toxicities.
  To evaluate the effect of maintenance therapy with decitabine on immune recovery including NK cells, Treg and Th17 T cells

CONTACTS AND LOCATIONS:
Overall Officials: Yoo-Jin Kim, MD, PhD, Principal Investigator — Division of Hematology,Department of Internal Medicine,Catholic Blood and Marrow Transplantation Center,Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Background] Bennett JM, Catovsky D, Daniel MT, Flandrin G, Galton DA, Gralnick HR, Sultan C. Proposals for the classification of the myelodysplastic syndromes. Br J Haematol. 1982 Jun;51(2):189-99. PMID 6952920
- [Background] Heaney ML, Golde DW. Myelodysplasia. N Engl J Med. 1999 May 27;340(21):1649-60. doi: 10.1056/NEJM199905273402107. No abstract available. PMID 10341278
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] Kolb HJ, Schattenberg A, Goldman JM, Hertenstein B, Jacobsen N, Arcese W, Ljungman P, Ferrant A, Verdonck L, Niederwieser D, van Rhee F, Mittermueller J, de Witte T, Holler E, Ansari H; European Group for Blood and Marrow Transplantation Working Party Chronic Leukemia. Graft-versus-leukemia effect of donor lymphocyte transfusions in marrow grafted patients. Blood. 1995 Sep 1;86(5):2041-50. PMID 7655033
- [Background] Cho BS, Kim YJ, Cho SG, Kim SY, Eom KS, Kim HJ, Lee S, Min CK, Kim DW, Lee JW, Min WS, Kim CC. The beneficial effect of chronic graft-versus-host disease on the clinical outcome of transplantation with fludarabine/busulfan-based reduced-intensity conditioning for patients with de novo myelodysplastic syndrome. Int J Hematol. 2007 Jun;85(5):446-55. doi: 10.1532/IJH97.A30616. PMID 17562624
- [Background] Kim YJ, Kim DW, Lee S, Min CK, Lee DG, Choi SM, Eom KS, Kim HJ, Lee JW, Min WS, Kim CC. Comparison of 2 preparative regimens for stem cell transplantation from HLA-matched sibling donors in patients with advanced myelodysplastic syndrome. Int J Hematol. 2005 Jul;82(1):66-71. doi: 10.1532/IJH97.A30501. PMID 16105763
- [Background] Kim SY, Cho SG, Cho BS, Kim MS, Eom KS, Kim YJ, Kim HJ, Lee S, Min CK, Kim DW, Lee JW, Min WS. Azacytidine treatment after discontinuation of immunosuppressants in patients with myelodysplastic syndrome and relapse after allo-SCT at a single center. Bone Marrow Transplant. 2010 Aug;45(8):1375-6. doi: 10.1038/bmt.2009.355. Epub 2009 Dec 21. No abstract available. PMID 20023706
- [Background] de Lima M, Giralt S, Thall PF, de Padua Silva L, Jones RB, Komanduri K, Braun TM, Nguyen HQ, Champlin R, Garcia-Manero G. Maintenance therapy with low-dose azacitidine after allogeneic hematopoietic stem cell transplantation for recurrent acute myelogenous leukemia or myelodysplastic syndrome: a dose and schedule finding study. Cancer. 2010 Dec 1;116(23):5420-31. doi: 10.1002/cncr.25500. Epub 2010 Jul 29. PMID 20672358
- [Derived] Han S, Kim YJ, Lee J, Jeon S, Hong T, Park GJ, Yoon JH, Yahng SA, Shin SH, Lee SE, Eom KS, Kim HJ, Min CK, Lee S, Yim DS. Model-based adaptive phase I trial design of post-transplant decitabine maintenance in myelodysplastic syndrome. J Hematol Oncol. 2015 Oct 23;8:118. doi: 10.1186/s13045-015-0208-3. PMID 26497198